CLINICAL TRIAL: NCT05129670
Title: Placebo Controlled, Confirmatory Clinical Investigation in Patients With Gastro-oesophageal Reflux, to Characterise the Acid Neutralisation Activity of a Calcite Chewing Gum, Using Oesophageal Ambulatory pH Monitoring
Brief Title: Clinical Investigation to Assess the Acid Neutralisation Activity of a Calcite Chewing Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5032701
Record Dates: First submitted 2021-10-26; First posted 2021-11-22 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2022-10

CONDITIONS: Esophagitis; Gastro Oesophageal Reflux Disease
Keywords: Gastro-oesophageal reflux disease
MeSH Terms: conditions — Esophagitis; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: This clinical investigation is being conducted to characterise the acid neutralisation activity of the test product, a calcite chewing gum, by comparing the antacid action with an unmatched placebo chewing gum. In this clinical investigation, the test product's ability to increase the pH within the oesophagus will be evaluated against an unmatched placebo.
Masking Description: Patients and the staff at the Investigative site, will remain un-masked to treatment administered. Masking of the investigation is not required as the investigation endpoints are objective measurements of oesophageal pH and impedance, patients will be randomised to a treatment order.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcite chewing gum (Experimental): Patients with a stable pH recording after fasting for at least 6 hours will receive a refluxogenic test meal which will be consumed within 30 mins. Thirty minutes after finishing the meal, the patient will be dosed with the randomised calcite chewing gum. pH and impedance measurements will be collected throughout the treatment period from the baseline assessment to 2 hours post dose
  Interventions: Device: Calcite chewing gum
- Unmatched Placebo chewing gum (Placebo Comparator): Patients with a stable pH recording after fasting for at least 6 hours will receive a refluxogenic test meal which will be consumed within 30 mins. Thirty minutes after finishing the meal, the patient will be dosed with the randomised unmatched placebo gum product. pH and impedance measurements will be collected throughout the treatment period from the baseline assessment to 2 hours post dose
  Interventions: Device: Unmatched Placebo chewing gum

INTERVENTIONS:
Device: Calcite chewing gum — The calcite chewing gum is administered as two pieces of gum in a single dose, 30 minutes following the consumption of a refluxogenic meal.
  Arms: Calcite chewing gum
Device: Unmatched Placebo chewing gum — The placebo chewing gum is administered as two pieces of gum in a single dose, 30 minutes following the consumption of a refluxogenic meal.
  Arms: Unmatched Placebo chewing gum

SUMMARY:
This investigation is designed to evaluate the acid neutralisation action of a new test product versus unmatched placebo.

DETAILED DESCRIPTION:
The primary objective of this confirmatory clinical investigation is to evaluate the acid neutralisation action of a calcite chewing gum, by comparing the antacid action with an unmatched placebo chewing gum. The clinical investigation will also assess the efficacy and safety of the calcite chewing gum.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a primary diagnosis of symptomatic GORD in accordance with the Montreal definition. Patients must have experienced frequent troublesome heartburn and / or regurgitation (with or without dyspepsia symptoms) of mild/moderate intensity. If the patient also has other symptoms, the heartburn, regurgitation or dyspepsia should be the predominant symptoms.
2. Patient that are healthy (with the exception of a diagnosis of GORD) as determined by past medical history and vital signs at screening.

Exclusion Criteria:

1. Patients with a history or active gastrointestinal disease (gastroduodenal ulcer, gastrointestinal haemorrhage, mechanical obstruction or perforation) or hiatus hernia which is greater than 3 cm or a history of conditions that can lead to abnormal oesophageal pH.
2. Patients experiencing frequent troublesome heartburn and / or regurgitation (with or without dyspepsia symptoms) of severe intensity
3. Patients who are unwilling to refrain from using antacids or alginates 24 hours prior to the start of the treatment visit.
4. Patients who are unwilling to refrain from using proton pump inhibitors (PPIs), H2 antagonists, motility stimulants or other medicines for relief of symptoms of acid reflux disease 2 weeks prior to the start of treatment period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
To measure efficacy of the calcite chewing gum versus unmatched placebo by measurement of the mean percentage of time (%) that the pH of the oesophagus is greater or equal to 4 up to 1 hour post dosing | 0 to 1 hour post dose
  The mean percentage of time (%) that pH is greater or equal to 4 within the oesophagus during the 0-1 hour post dose monitoring period.

SECONDARY OUTCOMES:
To evaluate the efficacy of the test product versus the unmatched placebo by measurement of the time (mins) taken to observe the first non-acidic reflux event (pH greater or equal to 4 throughout event) immediately after the start of dosing | 0 to 2 hours post dose
  Time (mins) to first non-acidic reflux event (pH greater or equal to 4 throughout event)
To evaluate the efficacy of the test product versus the unmatched placebo by recording the number of acid reflux events (pH is below pH 4) for up to 2 hours post dose | 0 to 2 hours post dose
  The number of acid reflux events (pH is below pH 4) for up to 2 hours post dose
To evaluate the efficacy of the test product versus the unmatched placebo by recording the total number of reflux events up to 2 hours post dose | 0 to 2 hours post dose
  The total number of reflux events for up to 2 hours post dose
To evaluate the efficacy of the test product versus the unmatched placebo by recording the mean percentage of time (%) that the pH within the oesophagus is raised greater or equal to 4 over the period 1-2 hour post dose | 1 to 2 hours post dose
  The mean percentage of time (%) that pH is greater or equal to 4 within the oesophagus during the 1-2 hour post dose monitoring period.
To evaluate the efficacy of the test product versus the unmatched placebo by recording the mean percentage of time (%) that the pH within the oesophagus is raised greater or equal to 4 over the period 0-2 hour post dose | 0 to 2 hours post dose
  The mean percentage of time (%) that pH is greater or equal to 4 within the oesophagus during the 0-2 hour post dose monitoring period.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Buckley, Dr, Principal Investigator — Mercy University Hospital
Locations (1):
- Mercy University Hospital, Cork, County Cork, Ireland

IPD SHARING:
Plan to Share IPD: No
IPD will be shared as per local regulations

REFERENCES:
- [Background] Vandenplas Y, Hassall E. Mechanisms of gastroesophageal reflux and gastroesophageal reflux disease. J Pediatr Gastroenterol Nutr. 2002 Aug;35(2):119-36. doi: 10.1097/00005176-200208000-00005. PMID 12187285
- [Background] DeMeester TR, Wang CI, Wernly JA, Pellegrini CA, Little AG, Klementschitsch P, Bermudez G, Johnson LF, Skinner DB. Technique, indications, and clinical use of 24 hour esophageal pH monitoring. J Thorac Cardiovasc Surg. 1980 May;79(5):656-70. PMID 7366233
- [Background] Hunt RH. Importance of pH control in the management of GERD. Arch Intern Med. 1999 Apr 12;159(7):649-57. doi: 10.1001/archinte.159.7.649. PMID 10218743